CLINICAL TRIAL: NCT05772585
Title: Characterization of Metabolomic Fingerprints in Patients With Acute Liver Failure and Acute-on-chronic Liver Failure With Hepatic Encephalopathy, and Influence of Liver Transplantation
Brief Title: Characterization of Metabolomic Fingerprints in Patients With Acute Liver Failure and Acute-on-chronic Liver Failure With Hepatic Encephalopathy
Acronym: EH-CASIMIR
Status: Withdrawn | Type: Observational
Why Stopped: competitor study
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221332
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Hepatic Encephalopathy; Acute Liver Failure; Acute on Chronic Liver Failure
Keywords: Hepatic Encephalopathy; Acute liver failure; Acute on chronic liver failure; Liver transplantation; Metabolomics
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Failure, Acute; Acute-On-Chronic Liver Failure | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients ALF and ACLF: patients with acute liver failure (ALF) and acute-on-chronic liver failure (ACLF) with hepatic encephalopathy
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — Blood collection (1 to 4 times for each patient) in order to perform metabolomic analyses of the plasmatic fingerprints of patients with hepatic encephalopathy
  Other Names: Metabolomics analyses, High resolution liquid phase mass spectrometry

SUMMARY:
Hepatic encephalopathy is a frequent complication of both acute liver failure (ALF) and acute-on-chronic liver failure (ACLF) and could be responsible among other neurological complications of residual impairment after liver transplantation. Specific metabolomic studies have shed light into pathophysiology. Nevertheless, whether HE metabolomic fingerprints differ between HE in ALF and HE in ACLF and their evolution after liver transplantation (LT) is unknown.

The aim of our study is to analyse the metabolomic fingerprint in plasma of 2 different groups of patients before and after LT:

* hospitalized patients with ALF and HE
* hospitalized patients with ACLF and HE We will analyse metabolomic results to explore if there is any difference in metabolomic fingerprints between these 2 groups and if LT modify the metabolomic fingerprint in plasma in these 2 groups and in the same way.

We will collect blood samples in these 2 groups on the day of HE occurring and then on day 1, day 7 and day 30 (+/- 2 days) after LT. We aim to enroll 10 patients in ALF group and 20 patients in ACLF group.

Inclusion criteria are defined as age > 18 years, patient presenting with ALF (Synthetic liver failure (INR > 1.5) with hepatic encephalopathy (grade 1-4 of West-Haven classification), without pre-existing hepatopathy, HE beginning within <26 weeks) or ACLF (≥ grade 1 from CANONIC criteria), and clinical HE (grade 1-4 of West-Haven classification) on the day of enrolment. Exclusion criteria are defined as age < 18 years, absence of HE, LT without pre-existing HE, patients who already undergone a LT, legally protected person.

An EDTA blood sample will be collected, centrifuged and frozen on the day of enrolment, then on day 1, day 7 and day 30 (+/- 2 days) after LT. Metabolomic analyses will be performed by different techniques but especially with high resolution liquid phase mass spectrometry in collaboration with CEA. Statistical analyses will be both univariate (Mann-Whitney or Wilcoxon tests) and multivariate (with a classical and adapted method for metabolomic studies: Partial Least-Squares Discriminant Analysis (PLS-DA)).

We expect to identify different metabolomic fingerprints between HE in both ALF and ACLF patients as well as different kinetics for symptoms resolution after LT. The long-term objective is to target the specific metabolic pathways for each group in order to allow development of new targeted drugs against HE in these 2 different conditions.

DETAILED DESCRIPTION:
Every patient admitted with hepatic encephalopathy and ALF or ACLF in Intensive Care Unit (ICU) or hepatology unit in both hospitals of Rennes University Hospital and La Pitié-Salpêtrière University Hospital will be screened by physicians for inclusion and exclusion criteria. If patients meet the criteria, their non-opposition of that of their next-of-kin (in case of disturbed neurological state) will be collected and an information paper will be given to them and their inclusion will be written in their medical file. On the same day (Day 0), a 6mL EDTA tube will be collected during a blood sample included in the standard patient care. Biological and demographic data collection will be done on day 0 too.

Then, patients will be followed-up during all the study duration and in case of LT, blood sample with 6mL EDTA tube will be collected on day 1, 7 and 30 after LT. Data collection will be performed at the time of each blood collection.

In case of the patient is not in hospital on the scheduled day, the blood collection will be performed on the very next outpatient consultation.

Every blood sample will be included as part of the blood samples for standard patient care and will under no circumstances be subject to a dedicated collection if the patient does not benefit from a test on the scheduled day.

If patient did not underwent LT during the follow-up, then only day 0 blood sample will be analyzed.

The blood samples will be centrifuged at 3000g for 10 min at 4°C, then the plasma will be collected and aliquoted in 4 Eppendorf with 400µL of plasma in each. All the aliquots will be stored at -80°C in the laboratories of the 2 centers.

After enrollment of the 30 expected patients, a secure transport network will be set up between the laboratories of the Rennes University Hospital and the Pitié-Salpêtrière University Hospital to the "Laboratoire d'Études du Métabolisme des Médicaments" of the CEA Saclay Center.

Processing and metabolomic analysis will be carried out in the CEA laboratory. These analyses will last approximately 2 weeks.

After having performed metabolites extraction in all the samples, high resolution liquid phase mass spectrometry will be done.

Finally, data analyses will be done with the CEA team and the manuscript will be written at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* patient presenting with:
* ALF (Synthetic liver failure (INR > 1.5) with hepatic encephalopathy (grade 1-4 of West-Haven classification), without pre-existing hepatopathy, HE beginning within <26 weeks)
* or ACLF (≥ grade 1 from CANONIC criteria)
* with clinical HE (grade 1-4 of West-Haven classification) on the day of enrolment

Exclusion Criteria:

* age < 18 years
* absence of HE
* LT without pre-existing HE
* patients who already undergone a LT
* other cause of neurological impairment
* Legally protected person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised for acute or acute-on-chronic liver failure, with hepatic encephalopathy and receiving a liver transplant following medical progression
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
comparison of metabolomic fingerprints of hepatic encephalopathy between ALF and ACLF | 6 months
  Partial Least-Squares Discriminant Analysis (PLS-DA).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas WEISS, MD, PhD, Principal Investigator — APHP

IPD SHARING:
Plan to Share IPD: No